CLINICAL TRIAL: NCT00060658
Title: Functional Neuroimaging of Calculus Problem Solving
Brief Title: Magnetic Resonance Imaging of Calculus Problem Solving
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030178; 03-N-0178
Record Dates: First submitted 2003-05-08; First posted 2003-05-09 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-03

CONDITIONS: Healthy
Keywords: Prefrontal Cortex; Calculation; Mathematician; Cognition; Brain Mapping; Healthy Volunteer; HV

SUMMARY:
This study will use magnetic resonance imaging (MRI) to identify brain regions involved in solving algebraic math problems. It will examine brain activation according to the level of difficulty and the number of steps required to solve the problem. This information will help identify a possible correlation between problem-solving strategies and patterns of brain activation.

Undergraduate or graduate students between 19 and 36 years of age who have completed at least 2 years of college, have had at least one college course in integral calculus, and who have no history of neurological disease may be eligible for this study. Candidates will be screened with a medical history, including psychiatric and neurological information.

Participants will be asked to mentally solve a variety of integral calculus problems while undergoing MRI scanning, a procedure that uses a strong magnetic field and radio waves to produce images of structural and chemical changes in the brain. During the scan, the subject lies on a table in a narrow cylinder (the scanner) containing a magnetic field. A problem and possible solution are presented to the subject, who presses a button to verify if the answer is correct. At the end of the test, the participant completes a follow-up questionnaire to determine the problem-solving strategies used.

DETAILED DESCRIPTION:
The purpose of this protocol is to localize the neural regions and systems mediating the forms of knowledge representations hypothesized by the principal investigator to be stored in the human prefontal cortex.

Utilizing experimental neuropsychological tasks during functional MRI on healthy, adult volunteers, we will investigate hypotheses regarding the role of the dorsolateral prefrontal cortex in mathematical cognition in a population of normal controls recruited among college and graduate students. We will also attempt to determine the relationship of mathematical cognition between non-frontal neural structures, such as left parietal lobe, and frontal neural structures involved in mechanistic plans, actions and mental sets.

The data collected will consist of behavioral measures of cognitive performance and corresponding fMRI images. The data that we collect in this protocol will be of value in identifying a set of neural regions and distributed networks mediating the forms of knowledge representation stored in the prefrontal cortex. We will also use the data obtained in these studies to constrain theories of frontal lobe function and to provide evidence for the role of specific frontal cortex sectors in specific cognitive functions.

ELIGIBILITY:
INCLUSION CRITERIA:

Graduate students and undergraduate students who have completed two years of college.

They also must have taken at least one college course in Integral Calculus.

Age range: 19-40.

Right-handedness (some left-handed subjects may be recruited for preliminary behavioral studies).

EXCLUSION CRITERIA:

Individuals with a neurological or psychiatric history or medical condition that would constrain interpretation of their performance during functional neuroimaging studies will be excluded.

Individuals with contraindications to exposure to high magnetic field.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 2003-05; Study Completion 2005-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States